CLINICAL TRIAL: NCT00349557
Title: Pilot Phase II Trial of Bevacizumab in Combination With Hormonal and Radiotherapy in Patients With High-Risk Prostate Cancer
Brief Title: Bevacizumab With Hormonal and Radiotherapy for High-Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI 3031500
Record Dates: First submitted 2006-07-05; First posted 2006-07-07 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; High-Risk Prostate Cancer; 1st line therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bevacizumab; bicalutamide; Goserelin; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Drug: bevacizumab, bicalutamide and goserelin
Procedure: intensity modulated radiation therapy (IMRT)

SUMMARY:
The purpose of this study is to determine the acute and late toxicities from radiation therapy in combination with bevacizumab (given every 2 weeks for 16 weeks then every 3 weeks for 12 weeks), bicalutamide (every day for 16 weeks) and goserelin (every 3 months for 2 years).

DETAILED DESCRIPTION:
Although there is no data on the toxicity with concurrent bevacizumab and hormonal therapy, the combination is not expected to increase toxicity seen when given as a single agent. Abnormal tumor microenvironments, tumor progression, and metastatic spread are major factors contributing to treatment failures in radiotherapy. Anti-VEGF agents (e.g. bevacizumab) can help overcome these factors through several different mechanisims.

Studies also demonstrate prolonged use of anti-VEGF agents with radiation therapy was more effective at preventing metastases from irradiated tumors compared to a short course. Patients generally start hormonal therapy and daily radiotherapy at the same time. This study will delay the start of radiotherapy until 8 weeks after the start of hormonal therapy and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* High Risk Prostate Cancer as defined as ONE of the following:

  1. Clinical T2b-T4
  2. Gleason sum score 8-10
  3. PSA more than 20 and Gleason sum score 7
  4. In addition, clinical T2a patients are eligible if 5 or more biopsies contain Gleason 4+3 cancer (minimum of 10 biopsies total required)
* No evidence of metastatic disease within 60 days of enrollment, confirmed by physical examination, chest x-ray, bone scan, and computed tomography of the abdomen and pelvis
* ECOG performance status of 0, 1 or 2

Exclusion Criteria:

* Concurrent or prior treatment with radiation, cytotoxic, biologic therapy for prostate cancer; any major surgery within four weeks, prior hormonal therapy (except finasteride for obstructive voiding symptoms)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study; Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Presence of central nervous system or brain metastases
* Blood pressure of >150/100 mmHg
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
To determine the acute (within 90 days from 1st day of radiation therapy) toxicities from intensity modulated radiation therapy (IMRT) in conjunction with bevacizumab, bicalutamide, and goserelin.

SECONDARY OUTCOMES:
To evaluate the late toxicities (>90 days from 1st day of radiation therapy) of IMRT, bevacizumab, bicalutamide, and goserelin. Patients will be followed on study for toxicity evaluation for at least one year from day 1 if radiation therapy.
To determine the tolerability of the combination of bevacizumab and hormonal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Vuky, MD, Principal Investigator — Virginia Mason Medical Center; Huong Pham, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States